CLINICAL TRIAL: NCT02578732
Title: BrUOG 318: FOLFOX-A For Locally Advanced Pancreatic Cancer: A Phase II Brown University Oncology Research Group Trial
Brief Title: FOLFOX-A For Locally Advanced Pancreatic Cancer: A Phase II Brown University Oncology Research Group Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 318
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Locally Advanced Pancreatic Cancer; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOXA (Experimental): Schema:
  1 cycle = 14 days **It will not be considered a deviation if a cycle or pre-cycle assessment must be adjusted to accommodate scheduling or holidays. Adjustment must be documented with reason to BrUOG**
  Abraxane ®: 150mg/m2 IV over 30 minutes, day 1 (administered first) every 14 days.
  Oxaliplatin: 85mg/m2, IV over 2 hours, day 1 every 14 days Leucovorin: 400mg/m2, IV over 2 hours, day 1 every 14 days 5-FU infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours.)
  * It is at the discretion of the treating physician to give Neulasta, 6 mg sq x 1 post treatment
  * Antiemetics will be administered as per standard institutional policy.
  Interventions: Drug: FOLFOXA

INTERVENTIONS:
Drug: FOLFOXA — Schema:
  1 cycle = 14 days **It will not be considered a deviation if a cycle or pre-cycle assessment must be adjusted to accommodate scheduling or holidays. Adjustment must be documented with reason to BrUOG**
  Abraxane ®: 150mg/m2 IV over 30 minutes, day 1 (administered first) every 14 days.
  Oxaliplatin: 85mg/m2, IV over 2 hours, day 1 every 14 days Leucovorin: 400mg/m2, IV over 2 hours, day 1 every 14 days 5-FU infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours.)
  * It is at the discretion of the treating physician to give Neulasta, 6 mg sq x 1 post treatment
  * Antiemetics will be administered as per standard institutional policy.
  Other Names: FOLFOXA is a combination treatment including: Abraxane, Oxaliplatin, Leucovorin

SUMMARY:
Preliminary data suggests that FOLFOX-A may have equal or superior activity as compared to FOLFIRINOX for patients with metastatic pancreatic cancer and appears to be better tolerated with the ability to administer at least 10 cycles of therapy. Investigators therefore will evaluate FOLFOX-A in a phase II study for patient with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
See summary above

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed pancreatic ductal adenocarcinoma. Patients with pathology or cytology showing carcinoma of pancreas or adenosquamous of the pancreas are also eligible.
* Locally advanced pancreatic cancer, including patients defined by Callery19 as "unresectable" and "borderline resectable" are eligible:
* Measurable disease as per RECIST 1.1
* No prior chemotherapy for pancreatic cancer.
* No major surgery within 3 weeks of the start of study treatment. Patients must have recovered from the side effects of any major surgery at the start of study treatment. For questions on if a surgery is deemed "major," definition by surgeon can be used for clarification. Laparoscopy and central venous catheter placement are not considered major surgery.
* No prior invasive malignancy within the prior two years. However, patients with an early stage malignancy that is not expected to require treatment in the next 2 years (such as early stage, resected breast cancer or asymptomatic prostate cancer) are eligible.
* ECOG performance status 0 or 1.
* Age ≥ 18
* Not pregnant and not nursing. Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to beginning of treatment. Post-menopausal women (surgical menopause or lack of menses >24 months) do not need to have a pregnancy test, please document status.
* Women of childbearing potential and sexually active males must use an effective contraception method 28 days prior to treatment, during treatment and for three months after completing treatment (men are to use contraception for six months post last dose of drug). Documentation of this being discussed required.
* Required Initial Laboratory Values:

  * Neutrophils ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions within 7 days prior to laboratory sample)
  * Hemoglobin > 9.0g/dL
  * Creatinine ≤ 1.5 mg/dL -or- creatinine clearance ≥ 60 mL/min
  * Total bilirubin <1. 5 x ULN
  * AST (SGOT) & ALT (SGPT) ≤ 2.5 x ULN
  * Alkaline phosphatase < 2.5xULN. (Patients with elevated alkaline phosphatase, total bilirubin, AST and ALT, who have subsequently undergone biliary stenting and their liver tests are improving, do not need to wait for their alkaline phosphatase to become < 2.5x ULN if their total bilirubin, AST and ALT have improved to within required study levels and the alkaline phosphatase is decreasing.)

Exclusion Criteria:

* Patients with metastatic disease
* Prior hypersensitivity to Oxaliplatin or Abraxane ® that in the investigators opinion would put the patient at risk if re-exposed
* Preexisting neuropathy is not allowed from any cause.
* Patients with serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive FOLFOX-A
* Patients with unstable biliary stents or with plastic stents. Information on type of stent is required at registration.
* Patients with active infection or fever (patients on antibiotics for infection or patients getting over a cold or seasonal virus are not excluded), or known historical or active infection with HIV, hepatitis B, or hepatitis C.
* Patients with active sepsis or pneumonitis.
* Patients with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies that in the investigator's opinion would put the patient at an increased risk.
* Uncontrolled diabetes. If patient has diabetes, confirmation on status (controlled or uncontrolled) required at registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — BrUOG
Locations (1):
- Rhode Island Hospital and The Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FOLFOXA
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOXA
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years] | 66 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of FOLFOX-A for Patients With Locally Advanced Pancreatic Cancer.
Time Frame: From date of start of treatment, until the date of first documented progression, whichever came first, assessed up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFOXA
Number analyzed (Participants) | 28
Participants
  Complete Response | 0
  Partial Response | 12
  Stable Disease | 12
  Progressive Disease | 4

2. Secondary Outcome: Overall Survival for Patients With Locally Advanced Pancreatic Cancer Treated With FOLFOX-A
Time Frame: During treatment (approximately every 2 weeks for up to 6 months), then approximately every 4 months for for a maximum of 5 years
Measure: Mean (Full Range); unit: months
Arm/Group | FOLFOXA
Number analyzed (Participants) | 28
months | 12.3 [2 to 36]

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 5 years. Adverse events were assessed until 30 days after the last dose of FOLFOX-A, up to 28 weeks
Arm/Group | FOLFOXA
All-Cause Mortality (participants affected / at risk) | 24/28
Serious Adverse Events (participants affected / at risk) | 8/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOXA (N=28)
Diarrhea (Gastrointestinal disorders) | 2
Depression (Psychiatric disorders) | 1
Fever (General disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Infection, other (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cardiac disorder, other (Cardiac disorders) | 1 — Takotsubo cardiomyopathy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOXA (N=28)
Neutropenia (Investigations) | 25
Thrombocytopenia (Investigations) | 17
Anemia (Blood and lymphatic system disorders) | 18
Peripheral sensory neuropathy (Nervous system disorders) | 25
Diarrhea (Gastrointestinal disorders) | 20
Anorexia (Metabolism and nutrition disorders) | 10
Vomiting (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 25
Mucositis oral (Gastrointestinal disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Weight loss (Investigations) | 19
Elevated AST/ALT (Investigations) | 12
Elevated alkaline phosphatase (Investigations) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT02578732/Prot_SAP_ICF_000.pdf